CLINICAL TRIAL: NCT01095926
Title: Phase II Pharmacokinetic Study to Assess the Age-dependency in the Clearance of Doxorubicin in Paediatric Patients With Solid Tumours and Leukaemia
Brief Title: Pharmacokinetic Study of Doxorubicin in Children With Cancer
Acronym: Doxo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC-MS-001; 2009-011454-17 (EudraCT Number)
Record Dates: First submitted 2010-03-22; First posted 2010-03-30 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2010-03

CONDITIONS: Wilms Tumor; Neuroblastoma; Soft Tissue Sarcoma; Acute Lymphoblastic Leukemia
Keywords: pharmacokinetic; doxorubicin; cancer; troponin; natriuretic peptide; cardiotoxicity; anthracyclines; Ewing; ALL
MeSH Terms: conditions — Wilms Tumor; Neuroblastoma; Sarcoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms; Cardiotoxicity | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxorubicin (Experimental)
  Interventions: Drug: doxorubicin

INTERVENTIONS:
Drug: doxorubicin — blood sampling before, during and after doxorubicin administration

SUMMARY:
Analyze pharmacokinetics of doxorubicin in children with cancer. Furthermore investigate the predictive role of troponin and natriuretic peptides for anthracycline-induced cardiotoxicity .

DETAILED DESCRIPTION:
* Paediatric patients up to the age of 17 years will be included. Number and time points of PK sampling will depend on age and tumour type.
* PK samples will be collected from two doxorubicin administrations. Analyzing samples from two doxorubicin administrations will allow distinguishing between interindividual, intraindividual and residual variability.
* Doxorubicin and its major metabolite doxorubicinol will be measured in plasma using HPLC
* In addition, the natriuretic peptide BNP and the precursors NT-pro ANP and NT-proBNP as well as troponin T will be measured in plasma up to 28 days after doxorubicin administration to evaluate their use as clinical markers for cardiotoxicity.
* A data set of max 5 samples (3 +2 (in the 1st + 2nd Doxorubicin sampling periods)) will be collected in the younger children (< 3 years) and a data set of max. 8 samples ( 5 + 3) will be collected in the older children. Samples will be taken at predefined time points/ time intervals.
* An additional DNA sample will be taken and analyzed for genetic polymorphisms. The influence of genotype on pharmacokinetics and metabolism will be investigated by appropriate statistical methods, including population pharmacokinetic analyses. Genes to study would include MDR1 and SLC22A16, both involved in the transport of doxorubicin and AKR1A1 and CBR1, both involved in the reduction of doxorubicin to doxorubicinol. Selected genotypes will be incorporated as covariates into the population pharmacokinetic models developed. The potential impact of genetic variation will be evaluated in the context of other sources of variability such as age, weight, gender etc

ELIGIBILITY:
Inclusion Criteria:

* patients ≤ 17 years of age
* plan to receive at least two cycles of doxorubicin
* must be enrolled in a national or European protocol for treatment of Wilms Tumours, Neuroblastoma, Soft tissue sarcoma, Ewing Sarcoma or Acute lymphoblastic leukaemia and must be treated with doxorubicin according to that protocol Or Patients < 3 years enrolled or listed in any national or European study protocol for any paediatric malignancy. Treatment with doxorubicin has to be according to that protocol.
* Parents or legal representative(s) must provide written informed consent to participate in the trial according to national regulations. Patients that are able to understand should provide assent to participate in the trial.
* Life expectancy of at least 3 month
* Karnofsky performance status of ≥ 70%
* Additional blood withdrawal is acceptable for the patient. The decision is left to the investigator

Exclusion Criteria:

* prior cardiac problems

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Assess age-dependency in pharmacokinetics of doxorubicin in paediatric patients with solid tumours and leukaemia | 24h
  Measure doxorubicin and doxorubicinol concentration in blood plasma. Collect samples at two different doxorubicin infusions.

SECONDARY OUTCOMES:
Assess interindividual, intraindividual and residual variability of PK parameters in children | 24h
  Measure doxorubicin and doxorubicinol concentration in blood plasma. Collect samples at two different doxorubicin infusions.
Assess relationship between PK parameters and patient characteristics | 24h
  Measure doxorubicin and doxorubicinol concentration in blood plasma. Collect samples at two different doxorubicin infusions.
Explore in a preliminary fashion genetic polymorphisms that may influence doxorubicin clearance | 5 years
  Obtain one whole blood sample per patient, if separate consent was given.
Evaluate the potential role of natriuretic peptides and troponin as indicators for subclinical cardiotoxicity | 1 month
  Measure troponin T, troponin I, BNP, NT-proBNP, NT-proANP. Collect samples at two different doxorubicin infusions before and up to 1month after doxorubicin administration.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Boos, MD, Prof., Study Chair — University Hospital Muenster
Locations (23):
- France (7):
  - Centre Oscar Lambret, Lille
  - CHU La Timone, Marseille
  - MD Nicolas Andre, National Study Manager France, Marseille
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Institut curie, Paris
  - Institut Gustanve Roussy, Paris
- Germany (6):
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Kiel, Kiel
  - Universitätsklinikum Münster, Münster
  - Klinikum Stuttgart, Stuttgart
- Italy (4):
  - Prof. Maurizio D'Incalci, National Study Manager Italy, Milan
  - Università degli Studi di Milano, Monza
  - Clinica di Oncoematologia Pediatrica, Padua
  - Università Cattolica di Roma, Rome
- United Kingdom (6):
  - Birmingham Childrens Hospital, Birmingham
  - St James's University Hospital, Leeds
  - Great Ormond Street Hospital for Children, London
  - Royal Manchester Childrens Hospital, Manchester
  - Prof. Alan Boddy, National Study Manager UK, Newcastle upon Tyne
  - Royal Victoria Infirmary, Sir James Spence Institute of Child Health, Newcastle upon Tyne